CLINICAL TRIAL: NCT06181357
Title: Randomized Trial Evaluating the Rate of Pneumothorax in Severe Emphysema Secondary to Endoscopic Volume Reduction With Two-stage ZEPHYR® Valves Versus Endoscopic Volume Reduction With One-stage ZEPHYR® Valves
Brief Title: Trial Evaluating the Rate of Pneumothorax in Severe Emphysema Secondary to Endoscopic Volume Reduction With Two-stage ZEPHYR® Valves Versus Endoscopic Volume Reduction With One-stage ZEPHYR® Valves
Acronym: REPEAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 87RI21_0031 (REPEAT)
Record Dates: First submitted 2023-12-04; First posted 2023-12-26 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: COPD
Keywords: Endobronchial Zephyr® valves; Endoscopic lung volume reduction; Pneumothorax; Emphysema; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pneumothorax; Emphysema | interventions — Pneumonectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- two-stage ZEPHYR® valves (Experimental)
  Interventions: Procedure: Endoscopic lung volume reduction in 2 stages
- one-stage ZEPHYR® valves (Sham Comparator)
  Interventions: Procedure: Endoscopic lung volume reduction in 1 stage

INTERVENTIONS:
Procedure: Endoscopic lung volume reduction in 2 stages — After the selection process, they will all be hospitalized in order to undergo an endoscopic lung volume reduction with Zephyr® valve under general anesthesia. In the experimental group, patients will be treated according to Limoges' treatment algorithm (2 stages)
  Arms: two-stage ZEPHYR® valves
Procedure: Endoscopic lung volume reduction in 1 stage — After the selection process, they will all be hospitalized in order to undergo an endoscopic lung volume reduction with Zephyr® valve under general anesthesia. In the control group, the entire lobe will be treated during one procedure
  Arms: one-stage ZEPHYR® valves

SUMMARY:
Chronic obstructive pulmonary disease (COPD) affects 3.5 million people and is the third leading cause of death worldwide. Emphysema involves air retention in the lungs and is ultimately responsible for a major deterioration in the quality of life. Available drug treatments have moderate efficacy whereas surgical lung volume reduction can improve exercise capacity when offered to a very selected population but at the cost of significant morbidity and mortality.

Endoscopic Lung Volume reduction with ZEPHYR® valves improves respiratory function at rest, exercise tolerance and quality of life in patients with little or no interlobar collateral ventilation.

If this technique has therefore proven its effectiveness, it is not devoid of complications and is notably responsible for pneumothorax in 27% of cases. The management of this complication is clearly codified, ranging from patient monitoring to the removal of one or more valves. It is therefore a subject of major concern for multiple reasons: high incidence, lengthening of hospital stay, increase in the overall cost of care, potential loss of benefit for the patient in the event of permanent withdrawal. valves and above all a potentially fatal event.

A new strategy for implanting ZEPHYR® valves in two stages has been developed in Limoges University Hospital. This innovative algorithm has been evaluated in several non-comparative single or multicenter studies. In those studies, pneumothorax' rate secondary to lung volume reduction with endobronchial valves is rated between 4.5 and 12%. The efficacy of the treatment appears to be comparable with the data found in the trials evaluating in which the entire lobe was treated in one procedure. Moreover, despite two procedures, there does not seem to be any increased risk of occurrence of other complications. Finally, the systematic scheduling of a thoracic computed tomography between the two procedures showed that 26.6% of patients presented a reduction in volume greater than 350mL despite incomplete treatment.

These data seem promising but no direct comparison with standard one-step treatment has ever been conducted so far.

DETAILED DESCRIPTION:
The Zephyr® valve was first implanted in 2001. Since then, 5 important studies have proven a clinical superiority compared to the existing standard of care. Bronchoscopic lung-volume reduction with the use of one-way endobronchial valves is a potential treatment for patients with severe emphysema. Loss of lung elastic recoil leads to airflow obstruction, gas trapping, and increased operating lung volumes. Lung volume reduction surgery (LVRS), resection of the most affected of the lung, has been clearly shown to improve outcomes in selected patient groups. The surgical intervention is, however, associated with significant morbidity and an early mortality rate of about 5%. Therefore, there is considerable interest in developing novel treatment approaches that can reduce lung volume and gas trapping, either more safely than LVRS or in patients for whom LVRS is not an option.

In the present study, 244 patients will be randomized. After the selection process, they will all be hospitalized in order to undergo an endoscopic lung volume reduction with Zephyr® valve under general anesthesia. Half of them, the experimental group, will be treated according to Limoges' treatment algorithm (2 stages). For the other half, the control group, the entire lobe will be treated during one procedure will. Both groups will receive the standard of care treatments, according to the Global initiative for chronic Obstructive Lung Disease recommendations (GOLD).

Both groups will be followed for one year:

* All the patients will undergo a thorax CT scan 45 days after implanting the last valve. Three follow-up consultations are planned at 45 days, 6, and 12 months. During these consultations, each patient will complete a Saint-George Respiratory Questionnaire (SGRQ) Test, a plethysmography and a 6-minutes walking test.
* Patients randomized in the experimental group will undergo a plethysmography and a thorax CT scan one day before the second procedure.

ELIGIBILITY:
Inclusion Criteria:

Patient able to give informed consent and participate in the study

* Age ≥ 35 years old and ≤ 80 years old at the time of signing the consent
* Emphysema (homogeneous or heterogeneous) on a recent CT scan (< 6 months). Heterogeneous emphysema defined by a difference of at least 15% destruction (threshold 910HU) between two adjacent lobes.
* Destruction ≥ 50% (threshold 910 HU) of the target lobe on the chest scanner
* Smoking quit for 3 months
* Dyspnea ≥ 2 according to the modified Medical Research Council (mMRC) questionnaire)
* Post-bronchodilator FEV between 15 and 50% theoretical
* Post-bronchodilator total lung capacity ≥ 100% theoretical and post-bronchodilator residual volume ≥ 175% theoretical
* Distance traveled during the TM6M ≥ 100m
* Member of or beneficiary of a social security scheme

Exclusion Criteria:

* Asthma considered as main diagnosis
* Recurrent exacerbations: (>3 over the last year or 2 requiring hospitalization)
* Myocardial infarction or stroke in the 6 months prior to inclusion
* Symptoms of heart failure in the 6 months prior to inclusion
* Chest CT abnormalities: giant bulla (occupying more than a third of the pulmonary field), paraseptal emphysema, pulmonary nodule greater than 0.8cm (not applicable pulmonary nodules known for more than a year and stable), fibrosing interstitial pneumonitis, dilated bronchi
* Pulmonary tomoscintigraphy:

  * Patients for whom the least perfused lobe is not the one with the highest emphysema destruction score
  * Patients with homogeneous emphysema for whom the perfusion delta (difference in perfusion between the ipsilateral lung and the treated lobe) is less than 10%
* Arterial blood gas analysis in ambient air: Hypoxemia in ambient air (PaO2 < 45 mmHg). Hypercapnia (PaCO2 > 55 mmHg)
* Echocardiography:

  * Left Ventricular Ejection Function < 45%
  * Systolic pulmonary arterial pressure > 45 mmHg
* History of pneumonectomy, lung surgery homolateral to the lobe targeted for endoscopic lung volume reduction
* History of pneumothorax homolateral to the lobe targeted for endoscopic lung volume reduction
* History of endoscopic volume reduction
* Oral corticosteroid therapy > 20 mg/day within the 4 weeks preceding inclusion
* Symptomatic bronchial dilatations, bronchial colonization with pseudomonas aeruginosa, multi-resistant bacteria or aspergillus origin
* Metastatic cancer undergoing treatment or whose treatments ended less than 5 years ago
* Pregnant or breastfeeding women
* Nickel allergy
* Patient under guardianship, curatorship or under judicial protection
* Participation in another interventional clinical research
* Any other condition which, in the opinion of the investigator, could interfere with the objective of the study or would cause the subject's participation in the study to be suboptimal, in particular (non-exhaustive list) unweaned alcoholism, substance abuse, non-compliance with usual follow-up visits)

secondary exclusion criteria:

- Evidence of collateral ventilation measured by the Chartis system

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2027-06-06 (Estimated); Study Completion 2027-06-06 (Estimated)

PRIMARY OUTCOMES:
Pneumothorax rate | 45 day
  Proportion of patients suffering from at least one pneumothorax rate between the beginning and the first 45 days following the end of lung volume reduction with ZEPHYR® valves

SECONDARY OUTCOMES:
Forced expiratory volume in one second (FEV1) measurement | 0 Day, 45 Day, 6 month and 12 month
  Functional parameters at rest (plethysmography) - assessment of FEV1 in liter
Force Vital Expiratory (FVE) measurement | 0 Day, 45 Day, 6 month and 12 month
  Functional parameters at rest (plethysmography) - assessment of FVE in Liter
Functional Residual Capacity (FRC) measurement | 0 Day, 45 Day, 6 month and 12 month
  Functional parameters at rest (plethysmography) - assessment of FRC in Liter
Inspiratory Capacity (IC) measurement | 0 Day, 45 Day, 6 month and 12 month
  Functional parameters at rest (plethysmography) - assessment of IC in Liter
Residual Volume (RV) measurement | 0 Day, 45 Day, 6 month and 12 month
  Functional parameters at rest (plethysmography) - assessment of RV in Liter
Residual Volume (RV) / Total Lung Capacity (TLC) ratio | 0 Day, 45 Day, 6 month and 12 month
  Functional parameters at rest (plethysmography) - assessment of ration RV/TLC in Liter
Exercise tolerance | 0 Day, 45 Day, 6 month and 12 month
  6 minutes walking test
Quality of life questionnaire | 0 Day, 45 Day, 6 month and 12 month
  EuroQol 5-Digit 5-level (EQ-5D-5L) questionnaire
Quality of life questionnaire | 0 Day, 45 Day, 6 month and 12 month
  COPD Assessment Test (CAT). Minimum score is 0 and maximum is 40
Quality of life questionnaire | 0 Day, 45 Day, 6 month and 12 month
  Saint-George Respiratory Questionnaire (SGRQ)
lobe volume reduction | 45 Day
  Target lobe volume reduction by Thorax scanner
Respiratory events | 12 month
  Study of morbidity and mortality. number of Respiratory events
Events related to the valves | 12 month
  Study of morbidity and mortality. number of events related to the valves
Revision bronchoscopies | 12 month
  Study of morbidity and mortality. Numbers of revision bronchoscopies
Death | 12 month
  Study of morbidity and mortality. numbers of death
responder's rate | 12 month
  In the experimental arm, responder's rate after the first procedure (despite infralobar treatment) defined by:
  * Plethysmography
    * FEV1: Improvement of equal or more than 12%
    * RV: Decrease of equal or more than 430mL
  * Thorax CT scan: target lobe volume reduction rated at more than 350mL.
Incremental Cost-Utility Ratio (ICUR) | 12 month
  Incremental Cost-Utility Ratio (ICUR) of the 2 intervention strategies expressed in euros per QALY gained in 12 months. The ICUR will be calculated on the basis of the following data:
  Quality of life assessed by the EQ-5D-5L questionnaire. Direct medical costs.

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - CHU de Bordeaux, Bordeaux
  - CHU de Brest, Brest
  - CHU de Dijon, Dijon
  - chu de Grenoble, Grenoble
  - CHU de Lille, Lille
  - CHU de Limoges, Limoges
  - APHM, Marseille
  - Hopital Saint Joseph, Marseille
  - CHU de Nice, Nice
  - APHP, Paris
  - CHU de Rouen, Rouen
  - chu de Strasbourg, Strasbourg
  - Hopital Foch, Suresnes
  - chu de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No